CLINICAL TRIAL: NCT04199026
Title: Pilot Trial of an Implantable Microdevice for In Vivo Drug Sensitivity Testing in Patients With Sarcomas
Brief Title: Implantable Microdevice for the Delivery of Drugs and Their Effect on Tumors in Patients With Metastatic or Recurrent Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-0171; NCI-2019-05820 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0171 (Other: M D Anderson Cancer Center); R01CA180279 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-12-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Sarcoma; Recurrent Sarcoma; Resectable Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Everolimus; ganitumab; Ifosfamide; Irinotecan; pazopanib; Polyethylene Glycols; polyethylene glycol 400; polyethylene glycol 8000; Temozolomide; temsirolimus; Sirolimus; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Feasibility (microdevice, surgery) (Experimental): Patients undergo percutaneous implantation of up to 3 drug delivery microdevices up to 2 days before standard of care surgery. Patients receive doxorubicin hydrochloride, ifosfamide, vincristine, irinotecan, temozolomide, pazopanib, everolimus, polyethylene glycol, ganitumab, and temsirolimus via the microdevice in the absence of unacceptable toxicity. At the time of surgery 2 days later, patients have the drug delivery microdevice(s) removed.
  Interventions: Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Device: Drug Delivery Microdevice; Drug: Everolimus; Biological: Ganitumab; Drug: Ifosfamide; Drug: Irinotecan; Drug: Pazopanib; Drug: Polyethylene Glycol; Drug: Temozolomide; Drug: Temsirolimus; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine

INTERVENTIONS:
Drug: Doxorubicin — Given via microdevice
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given via microdevice
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Device: Drug Delivery Microdevice — Undergo percutaneous implantation of drug delivery microdevice
  Other Names: Microdevice
Drug: Everolimus — Given via microdevice
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Biological: Ganitumab — Given via microdevice
  Other Names: AMG 479; Anti-IGF-1R Human Monoclonal Antibody AMG-479
Drug: Ifosfamide — Given via microdevice
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Irinotecan — Given via microdevice
Drug: Pazopanib — Given via microdevice
  Other Names: GW786034
Drug: Polyethylene Glycol — Given via microdevice
  Other Names: Glycol, polyethylene; PEG; Poly(oxyethylene); Polyethylene Glycol 400; Polyethylene Glycol 8000; POLYETHYLENE GLYCOL, UNSPECIFIED; Polyethylene Oxide
Drug: Temozolomide — Given via microdevice
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
Drug: Temsirolimus — Given via microdevice
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery
Drug: Vincristine — Given via microdevice
  Other Names: LEUROCRISTINE; VCR; Vincrystine

SUMMARY:
This early phase I trial studies the side effects of implanting and removing a microdevice in patients with sarcomas that have spread to other places in the body (metastatic) or have come back (recurrent). Microdevices are rice-sized devices that are implanted into tumor tissue and are loaded with 10 different drugs that are delivered at very small doses, or "microdoses," which may only affect a very small, local area inside the tumor. The purpose of this study is to determine which drugs delivered in the microdevice affect tumor tissue in patients with sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety of drug delivery microdevice (microdevice) placement and removal in subjects undergoing resection of sarcoma.

II. Determine the technical feasibility of microdevice placement and removal with intact surrounding tissue in subjects undergoing resection of a sarcoma.

SECONDARY OBJECTIVE:

I. Use the intratumoral cellular response to evaluate individual agents and/or drug combinations released from the microdevice reservoirs to assess the relative drug efficacy across all individual agents or drug combinations tested using the microdevice technology.

EXPLORATORY OBJECTIVES:

I. Evaluate the microdevice performance for its capacity to predict Response Evaluation Criteria in Solid Tumors (RECIST) response in the subset of patients that receive systemic chemotherapies as part of their standard-of-care or clinical trial treatments. II. Determine genomic, transcriptomic, and proteomic predictive biomarkers from resected specimens that correlate with local (i.e. microdevice-based) and systemic drug response. III. Determine, at a single-cell level, proteomic traits associated with chemosensitivity versus (vs.) resistance using mathematical notions of network robustness and fragility.

OUTLINE:

Patients undergo percutaneous implantation of up to 3 drug delivery microdevices up to 2 days before standard of care surgery. Patients receive doxorubicin hydrochloride, ifosfamide, vincristine, irinotecan, temozolomide, pazopanib, everolimus, polyethylene glycol, ganitumab, and temsirolimus via the microdevice in the absence of unacceptable toxicity. At the time of surgery 2 days later, patients have the drug delivery microdevice(s) removed. Conditions Conditions: Metastatic Sarcoma Recurrent Sarcoma

ELIGIBILITY:
Inclusion:

* Patients with a biopsy-confirmed recurrent or metastatic sarcoma for which surgery is indicated as a standard of care.
* 10 years of age or older
* Documented, signed, dated informed consent to participate in the microdevice study
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2

Exclusion:

* Subjects who do not wish to undergo surgical resection, or those who are high-risk or not candidates for surgical resection
* Age < 10 years old
* Women of childbearing potential without a negative pregnancy test; or women who are lactating
* Allergies or prior adverse drug reactions to any of the drugs loaded within the microdevice.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the safety and technical feasibility of microdevice insertion/removal, as assessed by adverse events by CTCAE 5.0. | Up to 1 year
  Assess the safety of microdevice placement and removal in subjects undergoing resection of sarcoma.
To assess efficacy across all individual agents or drug combinations tested using the microdevice technology. | Up to 1 year
  The primary outcome measure is the number of participants that experience a grade 3 or 4 adverse event, as defined by CTCAE 5.0. A second primary outcome measure of device technical feasibility measures the number of devices that successfully generate high-quality data from each of at least 50% of the patients enrolled. A successful device is one that generated high-quality data from at least 40% of the drugs in the device by IHC and/or other methodologies

SECONDARY OUTCOMES:
Determine the drug antineoplastic drug effects observed in the adjacent tumor tissues following exposure to drug micro-doses released by each microdevice reservoir. | Up to 1 year
  The degree of cell apoptosis and cell proliferation observed in the adjacent tumor tissues will be compared for the placebo control (i.e. PEG) to gauge the antineoplastic effect elicited by each of the drug micro-doses released by the respective microdevice reservoirs.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ludwig, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT04199026/ICF_000.pdf